CLINICAL TRIAL: NCT04638348
Title: A Novel Biofeedback Device to Improve Adherence to Pelvic Floor Muscle Training in Women With Urinary Incontinence: A Randomized Controlled Pilot Trial
Brief Title: A Novel Biofeedback for Urinary Incontinence in Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Kwong Wah Hospital (Other)
Responsible Party: Principal Investigator, Dr. Priya Kannan, Assistant Professor, The Hong Kong Polytechnic University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P0033900
Record Dates: First submitted 2020-11-16; First posted 2020-11-20 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Stress Urinary Incontinence
Keywords: Biofeedback
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- New Biofeedback (Experimental): Women allocated to the new biofeedback group will be instructed to attach the biofeedback device to their underpants and then perform pelvic floor muscle training.
  Interventions: Device: New Biofeedback
- Conventional Biofeedback (Active Comparator): Women allocated to the conventional biofeedback group will undergo pelvic floor muscle training with the conventional biofeedback probe inserted in the vagina
  Interventions: Device: New Biofeedback
- Control group (Active Comparator): The control group will perform pelvic floor muscle training without any biofeedback device.
  Interventions: Device: New Biofeedback

INTERVENTIONS:
Device: New Biofeedback — Conventional biofeedback consists of a electromyography biofeedback device with a vaginal probe.
  Other Names: Conventional Biofeedback

SUMMARY:
A three-armed randomized pilot trial will be conducted with 51 women having stress urinary incontinence, to evaluate the acceptance and ease of use of the conventional electromyography (EMG) biofeedback via vaginal probe in the treatment of urinary incontinence and that of the newly developed EMG biofeedback with Bluetooth. Women will be randomly allocated to one of two intervention groups (new biofeedback or conventional biofeedback) or the control group (PFMT alone). Women in the intervention groups will perform PFMT either with the new biofeedback or the conventional biofeedback, based on their group allocation. The control group will perform PFMT without a biofeedback device. Study outcome measures include, feasibility measures, International Consultation on Incontinence Questionnaire, and 1-hour pad test.

DETAILED DESCRIPTION:
Objectives: (1) to compare the acceptance and ease of use of the conventional electromyography (EMG) biofeedback via vaginal probe in the treatment of urinary incontinence and that of the newly developed EMG biofeedback with Bluetooth; (2) to investigate the effects of conventional biofeedback, the new biofeedback, and pelvic floor muscle training (PFMT) alone on urinary incontinence and adherence to PFMT.

Hypotheses: (1) The new biofeedback will be easier to use and women will more readily accept it than the conventional biofeedback. (2) Women assigned to the new biofeedback group will report better adherence to PFMT and greater improvements in urinary incontinence than women assigned to participate in the conventional biofeedback group.

Design and subjects: A three-armed randomized pilot trial will be conducted with 51 women who have stress urinary incontinence.

Interventions: Women will be randomly allocated to one of two intervention groups (new biofeedback or conventional biofeedback) or the control group (PFMT alone). Women in the intervention groups will perform PFMT either with the new biofeedback or the conventional biofeedback, based on their group allocation. The control group will perform PFMT without a biofeedback device.

Outcome measures: Feasibility measures, International Consultation on Incontinence Questionnaire, and 1-hour pad test.

Data analysis and expected results: A one-way between-groups analysis of covariance will be conducted. Adherence to PFMT will be better in the new biofeedback group than in the conventional biofeedback group. New biofeedback will have greater beneficial effects on urinary incontinence than either the conventional biofeedback or PFMT alone.

ELIGIBILITY:
Inclusion Criteria:

* women in the age group of 35 to 60 years of age;
* non-pregnant;
* having stress urinary incontinence;
* experiencing mild to moderate urinary incontinence (obtaining a score of ≤ 12 on the short-form of the International Consultation on Incontinence Questionnaire (ICIQ-sf); and
* obtaining a mini-mental state examination (MMSE) score of ≥ 24.

Exclusion Criteria:

* being in the postpartum stage of < 6 months;
* having severe pelvic organ prolapse (stages 3 and 4 on the Baden and Walker grading tool);
* women taking any medications that might cause urine retention;
* women having complicated UI due to radiation to pelvic region;
* obesity with a body mass index ≥ 30;
* women with incontinence secondary to other medical conditions or previous surgeries;
* women with severe psychological problems impairing participation in the study; and
* women having mixed or urge UI.

Ages: 35 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity as female
Enrollment: 51 (Actual)
Dates: Start 2020-02-01 (Actual); Primary Completion 2021-09-29 (Actual); Study Completion 2021-09-29 (Actual)

PRIMARY OUTCOMES:
Recruitment rate | At the end of recruitment period
  Number of participants recruited/screened in a week, the time taken for recruitment of participants, and reasons for declining to participate will be recorded.
Adherence | Post-intervention at 6 months
  The 0-10-point scale of the reliable tool (Cronbach's α=0.7059) developed to monitor long-term adherence to PFMT in women with UI (that quantifies adherence to home exercise as "low," "moderate," or "high") will be used to evaluate adherence to PFMT with and without the biofeedback device
Retention rate | Post-treatment at 1, 3 and 6 months
  This will be calculated as the percentage of participants who completed assessments at 1, 3, and 6 months.

SECONDARY OUTCOMES:
International Consultation on Incontinence Questionnaire-short form | Baseline (pre-intervention), post-treatment at 1, 3 and 6 months
  Measures amount of urine loss and intensity. Higher score indicates more sever urinary incontinence.
one-hour pad test with stress test | Baseline (pre-intervention), post-treatment at 1, 3 and 6 months
  Measure amount of urine leakage. Larger the amount of urine lost in grams, greater is the severity of urinary incontinence.
Modified Oxford scale | Baseline (pre-intervention), post-treatment at 1, 3 and 6 months
  To grade pelvic floor muscle strength. Lower the score, lower the strength of the pelvic floor muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Priya Kannan, PhD, Principal Investigator — The Hong Kong Polytechnic Unviersity
Locations (1):
- Kwong Wah Hospital, Kowloon, Hong Kong

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kannan P, Cheing GLY, Fung BKY, Li J, Leung WC, Chung RCK, Cheung TW, Lam LF, Lee WY, Wong WC, Wong WH, Tang PYG, Chan PKL. Effectiveness of pelvic floor muscle training alone or combined with either a novel biofeedback device or conventional biofeedback for improving stress urinary incontinence: A randomized controlled pilot trial. Contemp Clin Trials. 2022 Dec;123:106991. doi: 10.1016/j.cct.2022.106991. Epub 2022 Nov 2. PMID 36332826